CLINICAL TRIAL: NCT01124604
Title: Phase II Study of JNS024ER in Japanese Subjects With Chronic Pain Due to Osteoarthritis of the Knee or Low Back Pain
Brief Title: An Efficacy and Safety Study for Tapentadol Extended Release (JNS024ER) in Chronic Pain Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016999; JNS024ER-JPN-N21 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2010-04-22; First posted 2010-05-17 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Pain; Low Back Pain; Back Pain; Osteoarthritis, Knee
Keywords: Pain; Low Back Pain; Back Pain; Osteoarthritis, Knee; Tapentadol; Tapentadol Hydrochloride Extended Release
MeSH Terms: conditions — Pain; Low Back Pain; Back Pain; Osteoarthritis, Knee | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol Hydrochloride (Experimental)
  Interventions: Drug: Tapentadol Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tapentadol Hydrochloride — Tapentadol hydrochloride extended release (ER) tablets 25 to 250 milligram (mg) will be administered orally twice daily for 12 weeks. Dose will be adjusted as per Investigator's discretion.
  Arms: Tapentadol Hydrochloride
Drug: Placebo — Placebo matched to tapentadol hydrochloride ER tablets 25 to 250 mg will be administered orally twice daily for 12 weeks. Dose will be adjusted as per Investigator's discretion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and to explore the pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of tapentadol hydrochloride extended release (ER) tablets in Japanese participants with moderate to severe chronic pain due to osteoarthritis (disorder in which the joints become painful and stiff) of knee or low back pain.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), multi-center (when more than one hospital or medical school team works on a medical research study), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-control (participants are randomly assigned to a test treatment or to an identical-appearing treatment that does not contain the test drug), parallel-group (each group of participants will be treated at the same time) comparison study in participants with chronic pain due to osteoarthritis of knee or low back pain. The study duration will be of 14 weeks, which consists of a screening period of 1 week during which the participants will be evaluated for study eligibility, a treatment period of 12 weeks and a follow-up period of 1 week. The treatment period will consist of titration period (from the initiation of the study treatment to determination of the individual's maintenance dose) and maintenance period (from completion of the titration period to the completion of the treatment period). An optimal dose (maintenance dose) will be determined for each participant during the titration period and the treatment will be continued at the maintenance dose to assess the efficacy and safety. Tapentadol hydrochloride ER tablets 25 to 250 milligram or placebo will be administered orally twice daily. Efficacy and safety of the participants will primarily be evaluated by change from baseline in average pain intensity score based on 11-point Numerical Rating Scale (NRS) and Clinical Opiate Withdrawal Scale (COWS), respectively. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic pain due to osteoarthritis of knee or low back pain continuing for at least 12 weeks before informed consent
* Participants who did not achieve adequate analgesia (pain control) with routine treatment with an oral non-opioid analgesic (drug used to control pain) at its usual upper-limit dose or at an adequate fixed dose for at least 14 consecutive days during the 12 weeks before informed consent
* Participants who have not experienced treatment with conventional opioids, except for short term use of opioid analgesics for treatment of post-operative acute pain more than 30 days before consent or temporary use of codeine phosphate or dihydrocodeine phosphate for purposes other than pain relief (e.g. for antitussive) more than 2 days before informed consent
* Participants with average pain intensity score of greater than or equal to 5 on an 11-point Numerical Rating Scale (NRS) during 48 hours before informed consent and are considered requiring opioid treatment by the Investigator
* Participants who are able to visit the medical institutions throughout the study period

Exclusion Criteria:

* Participants who are taking a monoamine oxidase inhibitor within 14 days before informed consent
* Participants with current or a history of epilepsy or seizure disorders
* Participants suspected with intracranial hypertension (e.g. traumatic encephalopathy)
* Participants with uncontrolled or clinically significant arrhythmia (irregular heart rate)
* Participants with moderate to severe liver dysfunction or severe renal dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (19):
- Japan (19):
  - Aichi
  - Amagasaki
  - Chiba
  - Chikushi
  - Edogawa City
  - Fukuoka
  - Fukushima
  - Hiratsuka
  - Kawasaki
  - Kōtō City
  - Matsudo
  - Meguro City
  - Minatoku
  - Niigata
  - Osaka
  - Sagamihara
  - Shibuya City
  - Shinjuku-Ku
  - Toshima-Ku

RESULTS

PARTICIPANT FLOW:
Groups:
- Tapentadol Hydrochloride: Tapentadol hydrochloride extended release (ER) tablets 25 to 250 milligram (mg) were administered orally twice daily for 12 weeks. Dose was adjusted as per Investigator's discretion.
- Placebo: Placebo matched to tapentadol hydrochloride ER tablets 25 to 250 mg were administered orally twice daily for 12 weeks. Dose was adjusted as per Investigator's discretion.
Period: Overall Study
Arm/Group | Tapentadol Hydrochloride | Placebo
Started | 60 | 31
Completed | 45 | 29
Not Completed | 15 | 2
Not completed — Adverse Event | 10 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol Hydrochloride | Placebo | Total
Number analyzed (Participants) | 60 | 31 | 91
Age Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (15.54) | 68.1 (13.73) | 65.1 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 20 | 62
  Male | 18 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 11-point Numerical Rating Scale (NRS) at Week 12
Description: Participants were asked to assess the average pain intensity on a 11-point NRS ranging from 0 (no pain) to 10 (maximum pain imaginable) by selecting a number applicable to their pain on the scale. The mean pain intensity during the past 74 hours (3 days) was evaluated at Baseline and the mean pain intensity during the past 12 hours was evaluated at subsequent study visits.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS) included all the randomly assigned participants who received at least 1 dose of study drug and had post-randomization efficacy data. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Baseline | 6.9 (1.17) | 6.9 (1.12)
  Change at Week 12 | -3.0 (1.99) | -2.9 (2.22)
Statistical Analysis 1: Comparison: Tapentadol Hydrochloride vs Placebo; Test type: Superiority or Other; Least Square (LS) Mean Difference = -0.1, 95% CI [-1.04 to 0.80], Standard Error of Mean 0.46 — Test for no difference between treatments was derived from Analysis of covariance (ANCOVA) model with factors treatment, disease and Baseline pain intensity as covariate

2. Secondary Outcome: Change From Baseline in 11-point Numerical Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had post-randomization efficacy data. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Change at Week 1 | -0.6 (1.03) | -0.7 (1.08)
  Change at Week 2 | -1.1 (1.26) | -1.3 (1.55)
  Change at Week 3 | -1.5 (1.54) | -1.6 (1.59)
  Change at Week 4 | -1.9 (1.59) | -1.8 (1.71)
  Change at Week 5 | -2.4 (1.63) | -2.0 (1.71)
  Change at Week 6 | -2.7 (1.90) | -2.3 (1.82)
  Change at Week 7 | -2.7 (1.86) | -2.6 (2.01)
  Change at Week 8 | -2.8 (1.91) | -2.6 (2.08)
  Change at Week 9 | -2.9 (1.90) | -2.7 (2.12)
  Change at Week 10 | -2.9 (1.98) | -2.8 (2.25)
  Change at Week 11 | -3.0 (2.02) | -2.9 (2.25)

3. Secondary Outcome: Percentage of Participants With Response Based on 11-point Numerical Rating Scale (NRS)
Description: Percentage of participants with improvement in mean NRS score by greater than or equal to 30 percent or 50 percent in the last week from Baseline were considered as responders. Participants were asked to assess the average pain intensity on a 11-point NRS ranging from 0 (no pain) to 10 (maximum pain imaginable) by selecting a number applicable to their pain on the scale.
Time Frame: Week 12
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had post-randomization efficacy data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Percentage of participants
  Greater than or equal to 30 percent improvement | 55.0 (1.17) [41.61 to 67.88] | 61.3 (1.12) [42.19 to 78.15]
  Greater than or equal to 50 percent improvement | 40.0 [27.56 to 53.46] | 48.4 [30.15 to 66.94]

4. Secondary Outcome: Number of Participants With Categorical Scores on Patient's Global Impression of Change (PGIC) Scale
Description: The PGIC is a 7-point scale that requires the participants to assess how much their illness has improved or worsened relative to a Baseline state at the beginning of the intervention. The response options are 1 = very much improved, 2 = much improved, 3 = minimally improve, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Week 8, Week 12
Population: FAS included all participants who received study drug and had post-randomization efficacy data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 47 | 29
Participants
  Week 8; Very Much Improved (n = 47, 29) | 13 (1.17) [41.61 to 67.88] | 5 (1.12) [42.19 to 78.15]
  Week 8; Much Improved (n = 47, 29) | 17 [27.56 to 53.46] | 9 [30.15 to 66.94]
  Week 8; Minimally Improved (n = 47, 29) | 12 | 9
  Week 8; No Change (n = 47, 29) | 2 | 4
  Week 8; Minimally Worse (n = 47, 29) | 1 | 2
  Week 8; Much Worse (n = 47, 29) | 2 | 0
  Week 12; Very Much Improved (n = 45, 29) | 14 | 5
  Week 12; Much Improved (n = 45, 29) | 16 | 9
  Week 12; Minimally Improved (n = 45, 29) | 9 | 8
  Week 12; No Change (n = 45, 29) | 4 | 5
  Week 12 ; Minimally Worse (n = 45, 29) | 0 | 2
  Week 12; Much Worse (n = 45, 29) | 2 | 0

5. Secondary Outcome: Number of Participants With Response Based on Physician's Global Assessment Scale
Description: Physician's Global Assessment Scale assesses the therapeutic efficacy (effectiveness) of the study drug for pain control on a 2-point scale of "effective" and "not effective".
Time Frame: Week 8, Week 12
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 47 | 29
Participants
  Week 8; Effective (n=47, 29) | 41 | 24
  Week 8; Not effective (n=47, 29) | 6 | 5
  Week 12; Effective (n=45, 29) | 40 | 21
  Week 12; Not effective (n=45, 29) | 5 | 8

6. Secondary Outcome: Number of Participants With Presence of Pain Based on Brief Pain Inventory-Short Form (BPI-sf) Scale
Description: BPI-sf is a self-evaluated pain assessment form consisting of 15 items (item 1 - presence of pain, item 2 - pain location, items 3 to 6 - pain severity, item 7 - status of pain treatment, item 8 - efficacy of pain treatment, and items 9a to 9g - interference of pain with daily life). Item 1 for presence of pain assesses the question: "Do you have any pain today other than everyday kinds of pain?" on a 2-point scale of "yes" or "no".
Time Frame: Baseline, Week 12
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had post-randomization efficacy data. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Participants
  Baseline (n=60,31) | 46 (1.17) [41.61 to 67.88] | 25 (1.12) [42.19 to 78.15]
  Week 12 (n=45, 29) | 25 | 21

7. Secondary Outcome: Number of Participants With 50 Percent Pain Relief Based on Brief Pain Inventory-Short Form (BPI-sf) Scale
Description: BPI-sf is a self-evaluated pain assessment form consisting of 15 items (item 1 - presence of pain, item 2 - pain location, items 3 to 6 - pain severity, item 7 - status of pain treatment, item 8 - efficacy of pain treatment, and items 9a to 9g - interference of pain with daily life). Item 8 for efficacy of pain treatment assesses number of participants with at least 50 percent pain relief during the last 24 hours on a scale ranging from 0 percent (no relief) to 100 percent (complete relief).
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Participants
  Baseline (n=60, 31) | 9 (1.17) [41.61 to 67.88] | 7 (1.12) [42.19 to 78.15]
  Week 12 (n=45, 29) | 10 | 4

8. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Total Score at Week 12
Description: BPI-sf consists of 15 items (item 1 - presence of pain, item 2 - pain location, items 3 to 6 - pain severity, item 7 - status of pain treatment, item 8 - efficacy of pain treatment, and items 9a to 9g - interference of pain with daily life). Total score is defined as the mean scores from items 3, 4, 5, 6 and 9 recorded on an 11-point scale where 0 = no pain and 10 = pain as bad as you can imagine. Negative change indicates an improvement in pain.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Total Score; Baseline (n=60, 31) | 5.4 (1.63) | 5.7 (1.36)
  Total Score; Change at Week 12 (n=45, 29) | -2.4 (2.01) | -2.3 (2.11)

9. Secondary Outcome: Change From Baseline in Sleep Latency Based on Sleep Questionnaire at Week 12
Description: Sleep Latency was addressed by the question: "How long after bedtime/lights out did you fall asleep last night?" and the change from Baseline in sleep latency was reported. Decrease in time indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had post-randomization efficacy data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 45 | 29
Minutes | 1.0 (41.06) | 1.2 (31.20)

10. Secondary Outcome: Change From Baseline in Time Slept Based on Sleep Questionnaire at Week 12
Description: Time slept was addressed by the question: "How long did you sleep last night?" and the change from Baseline in time slept was reported.
Time Frame: Baseline, Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 45 | 29
Hours | 0.1 (1.50) | 0.2 (1.04)

11. Secondary Outcome: Number of Participants With Awakenings Based on Sleep Questionnaire
Description: Number of awakenings was addressed by the question: "How many times did you wake up during the night?'' and lesser number signified better sleep.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Participants
  Baseline; 0 awakening (n=60,31) | 10 [41.61 to 67.88] | 6 [42.19 to 78.15]
  Baseline; 1 awakening (n=60,31) | 18 (1.55) | 6 (1.00)
  Baseline; 2 awakenings (n=60,31) | 16 | 10
  Baseline; 3 awakenings (n=60,31) | 10 | 7
  Baseline; 4 awakenings (n=60,31) | 2 | 1
  Baseline; >= 5 awakenings (n=60,31) | 4 | 1
  Week 12; 0 awakening (n=45,29) | 9 | 6
  Week 12; 1 awakening (n=45,29) | 20 | 9
  Week 12; 2 awakenings (n=45,29) | 9 | 6
  Week 12; 3 awakenings (n=45,29) | 3 | 7
  Week 12; 4 awakenings (n=45,29) | 2 | 1
  Week 12; >=5 awakenings (n=45,29) | 2 | 0

12. Secondary Outcome: Number of Participants With Response Based on Overall Quality of Sleep Questionnaire
Description: Overall quality of sleep was addressed by the question: "Please rate the overall quality of your sleep last night" and participants could choose one of the following options: excellent, good, fair or poor.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Participants
  Baseline; Excellent (n=60, 31) | 1 [41.61 to 67.88] | 1 [42.19 to 78.15]
  Baseline; Good (n=60, 31) | 37 (1.55) | 17 (1.00)
  Baseline; Fair (n=60, 31) | 19 | 13
  Baseline; Poor (n=60, 31) | 3 | 0
  Week 12; Excellent (n=45, 29) | 2 | 0
  Week 12; Good (n=45, 29) | 30 | 21
  Week 12; Fair (n=45, 29) | 9 | 7
  Week 12; Poor (n=45, 29) | 4 | 1

13. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey Version 2 (SF-36v2) Scores at Week 12
Description: SF-36v2 is 36-item form related to 8 health concepts (physical functioning, role physical, role emotional, general health, social functioning, bodily pain, vitality, mental health) and 2 summary scores (physical and mental component summary). Physical functioning, role physical and bodily pain contribute to physical component; role emotional, social functioning and mental health contribute to mental component; and social functioning, vitality, and general health contribute to both. All scores are based on a scale from 0 to 100, with higher scores defining more favorable health state.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Physical Functioning; Baseline (n=60, 31) | 48.9 (18.18) [41.61 to 67.88] | 51.9 (24.65) [42.19 to 78.15]
  Physical Functioning; Change at Week 12 (n=45, 29) | 12.1 (18.01) | 3.4 (16.26)
  Role-Physical; Baseline (n=60, 31) | 57.8 (27.46) | 57.1 (26.41)
  Role-Physical; Change at Week 12 (n=45, 29) | 9.6 (30.05) | -0.4 (32.13)
  Bodily Pain; Baseline (n=60, 31) | 34.7 (15.53) | 34.3 (14.80)
  Bodily Pain; Change at Week 12 (n=45, 29) | 19.4 (20.91) | 15.1 (19.89)
  General Health; Baseline (n=60, 31) | 47.6 (15.14) | 47.8 (18.13)
  General Health; Change at Week 12 (n=45, 29) | 9.1 (13.81) | 4.7 (14.18)
  Vitality; Baseline (n=60, 31) | 46.4 (21.54) | 51.4 (16.67)
  Vitality; Change at Week 12 (n=45, 29) | 7.6 (16.20) | 3.7 (17.56)
  Social Functioning; Baseline (n=60, 31) | 66.5 (26.29) | 66.1 (23.09)
  Social Functioning; Change at Week 12 (n=45, 29) | 12.5 (21.65) | 5.2 (32.13)
  Role-Emotional; Baseline (n=60, 31) | 63.6 (28.29) | 61.0 (28.25)
  Role-Emotional; Change at Week 12 (n=45, 29) | 10.7 (25.23) | 2.6 (31.58)
  Mental Health; Baseline (n=60, 31) | 58.7 (22.17) | 59.7 (20.08)
  Mental Health; Change at Week 12 (n=45, 29) | 7.4 (20.16) | 6.4 (19.08)
  Mental Summary; Baseline (n=60, 31) | 47.5 (10.60) | 48.6 (9.99)
  Mental Summary; Change at Week 12 (n=45, 29) | 3.6 (7.49) | 3.6 (8.71)
  Physical Summary; Baseline (n=60, 31) | 25.5 (13.60) | 25.2 (16.75)
  Physical Summary; Change at Week 12 (n=45, 29) | 7.9 (12.78) | 1.3 (15.76)

14. Secondary Outcome: Change From Baseline in Western Ontario MacMaster Questionnaire (WOMAC) Global Score at Week 12
Description: WOMAC is a self administered 24-item questionnaire used to evaluate participants with osteoarthritis of the knee. It consists of 3 subscales: pain (5 items), joint stiffness (2 items), and physical function (17 items). Each item is assessed on a 5-point scale from 0 to 4. The global score assesses pain, disability and joint stiffness and ranges from 0 to 96. Higher scores indicate that a symptom is bothersome and physically disabling.
Time Frame: Baseline, Week 12
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had post-randomization efficacy data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 27 | 13
Units on a scale
  Global Score; Baseline (n=27, 13) | 1.9 (0.64) | 1.7 (0.64)
  Global Score; Change at Week 12 (n=20, 13) | -0.9 (0.56) | -0.4 (0.66)

15. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RDQ) Score at Week 12
Description: RDQ scale is used to assess the impact of low back pain on daily activities by participants. The scale consists of 24 item questionnaire with options as "Yes"/"No" where "Yes" is counted as 1 point. The total score ranged from 0 to 24, with higher scores indicating greater disability.
Time Frame: Baseline, Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 33 | 18
Units on a scale
  Baseline (n=33, 18) | 11.7 (5.08) | 12.7 (5.35)
  Change at Week 12 (n=25, 16) | -3.3 (4.25) | -1.8 (3.04)

16. Other Pre Specified Outcome: Number of Participants With Response Based on Clinical Opioid Withdrawal Symptoms Questionnaire (COWS)
Description: COWS is an 11-item questionnaire for clinical assessment of withdrawal symptoms. Total score is calculated by adding the scores of all the 11-items. The severity of withdrawal symptoms is categorized using values of total score as: 0-4 = no withdrawal, 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, and 37-48 = severe withdrawal.
Time Frame: Week 12
Population: Safety population included all the participants who received at least 1 dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Tapentadol Hydrochloride | Placebo
Number analyzed (Participants) | 60 | 31
Participants
  No Withdrawal | 60 (1.17) [41.61 to 67.88] | 31 (1.12) [42.19 to 78.15]
  Mild | 0 | 0
  Moderate | 0 | 0
  Moderately Severe | 0 | 0
  Severe Withdrawal | 0 | 0

17. Other Pre Specified Outcome: Serum Concentration of Tapentadol
Time Frame: Week 2, 4, 8, 12
Population: Pharmacokinetic analysis set included all participants who received at least 1 dose of study drug and had at least 1 serum study drug concentration. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tapentadol Hydrochloride
Number analyzed (Participants) | 60
nanogram per milliliter
  Tapentadol Hydrochloride 25 mg Week 2, n=11 | 14.1 (6.02)
  Tapentadol Hydrochloride 50 mg Week 2, n=48 | 29.7 (17.1)
  Tapentadol Hydrochloride 100 mg Week 2, n=1 | 47.9 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at given time point.
  Tapentadol Hydrochloride 150 mg Week 2, n=0 | NA (NA) — Data was not analyzed as no participant was evaluable for this dose at given time point.
  Tapentadol Hydrochloride 200 mg Week 2, n=0 | NA (NA) — Data was not analyzed as no participant was evaluable for this dose at given time point.
  Tapentadol Hydrochloride 250 mg Week 2, n=0 | NA (NA) — Data was not analyzed as no participant was evaluable for this dose at given time point.
  Tapentadol Hydrochloride 25 mg Week 4, n=4 | 22.8 (11.6)
  Tapentadol Hydrochloride 50 mg Week 4, n=10 | 23.6 (6.20)
  Tapentadol Hydrochloride 100 mg Week 4, n=28 | 59.0 (42.7)
  Tapentadol Hydrochloride 150 mg Week 4, n=16 | 76.2 (48.5)
  Tapentadol Hydrochloride 200 mg Week 4, n=0 | NA (NA) — Data was not analyzed as no participant was evaluable for this dose at given time point.
  Tapentadol Hydrochloride 250 mg Week 4, n=0 | NA (NA) — Data was not analyzed as no participant was evaluable for this dose at given time point.
  Tapentadol Hydrochloride 25 mg Week 8, n=3 | 25.1 (15.3)
  Tapentadol Hydrochloride 50 mg Week 8, n=8 | 22.7 (12.2)
  Tapentadol Hydrochloride 100 mg Week 8, n=16 | 57.7 (40.7)
  Tapentadol Hydrochloride 150 mg Week 8, n=13 | 83.2 (35.9)
  Tapentadol Hydrochloride 200 mg Week 8, n=4 | 87.8 (58.9)
  Tapentadol Hydrochloride 250 mg Week 8, n=4 | 147 (119)
  Tapentadol Hydrochloride 25 mg Week 12, n=3 | 29.2 (13.2)
  Tapentadol Hydrochloride 50 mg Week 12, n=8 | 25.1 (8.17)
  Tapentadol Hydrochloride 100 mg Week 12, n=14 | 49.1 (36.3)
  Tapentadol Hydrochloride 150 mg Week 12, n=12 | 40.4 (33.9)
  Tapentadol Hydrochloride 200 mg Week 12, n=4 | 119 (165)
  Tapentadol Hydrochloride 250 mg Week 12, n=4 | 130 (77.6)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days post last study dose
Arm/Group | Tapentadol Hydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 3/60 | 0/31
Other Adverse Events (participants affected / at risk) | 54/60 | 24/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Hydrochloride (N=60) | Placebo (N=31)
Aortic dissection (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Hydrochloride (N=60) | Placebo (N=31)
Nasopharyngitis (Infections and infestations) | 14 | 2
Cystitis (Infections and infestations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 7 | 0
Somnolence (Nervous system disorders) | 22 | 3
Dizziness (Nervous system disorders) | 5 | 2
Headache (Nervous system disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 20 | 5
Constipation (Gastrointestinal disorders) | 13 | 2
Vomiting (Gastrointestinal disorders) | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Renal impairment (Renal and urinary disorders) | 2 | 2
Thirst (General disorders) | 6 | 2
Drug withdrawal syndrome (General disorders) | 6 | 0
Malaise (General disorders) | 5 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 2
Blood pressure increased (Investigations) | 1 | 2
Blood triglycerides increased (Investigations) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 0
Thermal burn (Injury, poisoning and procedural complications) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Feeling abnormal (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Face oedema (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood urea increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood urine present (Investigations) | 1 | 1
White blood cell count increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0
Respiratory rate increased (Investigations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Vascular insufficiency (Vascular disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.